CLINICAL TRIAL: NCT01367925
Title: A Prospective, Randomized, Comparison of Total Knee Arthroplasty With the Triathlon® CS Tibial Insert vs. the Triathlon® PS Tibial Insert.
Brief Title: Stryker Triathlon® Cruciate Substituting vs. Posterior Stabilized Outcomes Study
Status: Completed | Type: Observational
Sponsor: Spokane Joint Replacement Center (Other)
Responsible Party: Principal Investigator, David F. Scott, MD, PI, Spokane Joint Replacement Center
Other Study IDs: SJRC-CS/PS
Record Dates: First submitted 2011-05-22; First posted 2011-06-07 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Total Knee Replacement; TKA; Knee; PS; CS
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cruciate Substituting Tibial Insert
  Interventions: Device: Stryker Triathlon® CS Tibial Insert
- Posterior Stabilized Tibial Insert
  Interventions: Device: Stryker Triathlon® PS Tibial Insert

INTERVENTIONS:
Device: Stryker Triathlon® CS Tibial Insert
  Groups: Cruciate Substituting Tibial Insert
Device: Stryker Triathlon® PS Tibial Insert
  Groups: Posterior Stabilized Tibial Insert

SUMMARY:
This study compares the clinical and radiographic outcomes obtained with the use of the Stryker Triathalon® Cruciate Substituting (CS) and Posterior Stabilized (PS) tibial inserts.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 20-80 years old
* Body mass index <40
* Undergoing primary total knee arthroplasty for osteoarthritis of the knee

Exclusion Criteria:

* Inflammatory arthritis
* Revisions

Other criteria may apply

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing total knee arthroplasty
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2007-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Clinical outcomes, Knee Society Score | Pre-operative, 6 weeks, 6 months, 1, 2, 3, 4, and 5 years post-operative
  Clinical outcomes to include overall success, failure rate, revison rate, clinical scores (Knee Society Score), range of motion, pain, stability, radiographic success

CONTACTS AND LOCATIONS:
Overall Officials: David F Scott, MD, Principal Investigator — Spokane Joint Replacement Center
Locations (1):
- Spokane Joint Replacement Center, Spokane, Washington, United States